CLINICAL TRIAL: NCT02143882
Title: A Phase III/IV Open-label Study of the Immunogenicity and Safety of a Single Dose of a Live Attenuated Influenza Vaccine (LAIV) (FluenzTM) for Each of Three Successive Years in Children naïve to, or in Previous Receipt of the AS03B Adjuvanted H1N1 (2009) Influenza Vaccine (Pandemrix ™).A Phase III/IV Open-label Study of the Immunogenicity and Safety of a Single Dose of a Live Attenuated Influenza Vaccine (LAIV) (FluenzTM) for Each of Three Successive Years in Children naïve to, or in Previous Receipt of the AS03B Adjuvanted H1N1 (2009) Influenza Vaccine (Pandemrix ™).
Brief Title: A Phase III/IV Open-label Study of the Immunogenicity and Safety of a Single Dose of a Live Attenuated Influenza Vaccine (LAIV) (FluenzTM) for Each of Three Successive Years in Children naïve to, or in Previous Receipt of the AS03B Adjuvanted H1N1 (2009) Influenza Vaccine (Pandemrix ™).
Acronym: LAIV Immuno
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: Institute of Child Health (Other)
Responsible Party: Principal Investigator, Prof. Elizabeth Miller, Consultant Epidemiologist, Public Health England
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAIV Immuno
Record Dates: First submitted 2014-05-13; First posted 2014-05-21 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Live Attenuated Influenza Vaccine
Keywords: Live attenuated influenza vaccine; fluenz; pandemrix; pandemic influenza vaccine; immunogenicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAIV (Experimental): All children will receive LAIV, currently available as the marketed product Fluenz
  Interventions: Drug: Fluenz

INTERVENTIONS:
Drug: Fluenz — Live attenuated influenza vaccine

SUMMARY:
The Department of Health has recently announced the implementation of annual vaccination for all those aged 18 years and under, with live attenuated influenza vaccine (LAIV), which is delivered as a nasal spray. This study seeks primarily to measure antibody responses to the LAIV vaccination over three subsequent years and will involve six blood samples, six dried blood spots (taken from the end of the blood sample needle) and six oral fluid samples - before and three weeks after each vaccination each year. These samples will allow us to assess how the immune system responds to the vaccinations in terms of the antibodies that are present.

DETAILED DESCRIPTION:
The Department of Health has recently announced the implementation of annual vaccination for all those aged 18 years and under, with live attenuated influenza vaccine (LAIV), which is delivered as a nasal spray. The programme will begin in the influenza season, from September 2013, with children aged 24 years of age, and older children being included from the influenza season of 2014. Therefore this study seeks primarily to measure antibody responses to the LAIV vaccination over three subsequent years and will involve six blood samples, six dried blood spots (taken from the end of the blood sample needle) and six oral fluid samples - before and three weeks after each vaccination each year. These samples will allow us to assess how the immune system responds to the vaccinations in terms of the antibodies that are present.

The study will specifically recruit children in previous receipt of Pandemrix, a pandemic influenza vaccine, and those naïve to pandemic influenza vaccination, which will allow the comparison of responses to LAIV between these groups.

The sample size required to answer the primary objective of the study is 200 evaluable children per group. As the study will be conducted over three years the recruitment target will be 500 children across the two groups to allow for the expected attrition of numbers over time.

The investigators will also be assessing how well the vaccines are tolerated and each participant will therefore be asked to complete a health diary for the week following vaccination. They will be asked to record any symptoms, which the investigators will elicit in line with the information in the Summary of Product Characteristics (SPC) as well as any illnesses or visits to their GP or hospital.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian gives written informed consent for participation of their child in the study.

  * Male or female aged 4 years (+364 days) to 8 years (+364 days) on the day of consent.
  * Documented prior receipt of Pandemrix, or no evidence in the medical notes of never having had pandemic influenza vaccine.

Exclusion Criteria:

* Absolute exclusion criteria. The participant may not enter the study if ANY of the following apply:

From Fluenz Summary of Product Characteristics (SPC):

* Hypersensitivity to the active substances, to any of the excipients (e.g. gelatin; see appendix 1), to gentamicin (a possible trace residue), to eggs or to egg proteins (e.g. ovalbumin).
* Children and adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and highdose corticosteroids. FLUENZ is not contraindicated for use in individuals with asymptomatic HIV infection; or individuals who are receiving topical/inhaled corticosteroids or lowdose systemic corticosteroids or those receiving corticosteroids as replacement therapy, e.g. for adrenal insufficiency.
* Children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wildtype influenza infection.

Study specific exclusions:

* Any contraindication to vaccination as specified in the "Green Book"Immunisation against Infectious Disease, HMSO.
* known bleeding diathesis (or any condition that may be associated with a prolonged bleeding time).
* Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study. *Temporary Exclusion Criteria

From the SPC:

• The concurrent use of FLUENZ with antiviral agents that are active against influenza A and/or B viruses has not been evaluated. However, based upon the potential for influenza antiviral agents to reduce the effectiveness of FLUENZ, it is recommended not to administer the vaccine until 48 hours after the cessation of influenza antiviral therapy.

Administration of influenza antiviral agents within two weeks of vaccination may affect the response of the vaccine.

Because of this information in the SPC, should any child be given these medications the administration of LAIV would be delayed as specified.

Study specific:

* Fever (sublingual temperature ≥ 38°C)
* Received any blood or blood products within the past 12 weeks.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Immune responses to LAIV | three subsequent years, all children
  To compare the immune response to homologous and heterologous strains before and after to annual doses of LAIV over three consecutive years in children aged 49(+364days) years at enrollment in naïve children vs those in previous receipt of the AS03B adjuvanted pandemic influenza vaccine to homologous vaccine strains .

SECONDARY OUTCOMES:
Incidence of influenza | all children, three subsequent years
  To document the incidence of laboratory confirmed influenza and other respiratory viruses in the naïve and Pandemrix™ primed children over the three seasons.
safety and tolerability of LAIV | all children, three years of participation
  To compare the safety and tolerability of annual doses of LAIV in naïve compared to Panemrix™ vaccinated children in terms of local and systemic reactions following vaccination as recorded in a health diary for the week following vaccination as well as any serious adverse events identified throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, Principal Investigator — Public Health England
Locations (2):
- United Kingdom (2):
  - Gloucestershire, Gloucestershire, Gloucestershire
  - Hertfordshire, Hertfordshire, Hertfordshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jackson D, Pitcher M, Hudson C, Andrews N, Southern J, Ellis J, Hoschler K, Pebody R, Turner PJ, Miller E, Zambon M. Viral Shedding in Recipients of Live Attenuated Influenza Vaccine in the 2016-2017 and 2017-2018 Influenza Seasons in the United Kingdom. Clin Infect Dis. 2020 Jun 10;70(12):2505-2513. doi: 10.1093/cid/ciz719. PMID 31642899
- See also: PHE website — https://www.gov.uk/government/organisations/public-health-england